CLINICAL TRIAL: NCT00003091
Title: Treatment of Metastatic Renal Cell Carcinoma and Melanoma With Subsequential High-Dose Subcutaneous Interferon Alfa-2b and High-Dose Bolus and Continuous Intravenous Interleukin-2
Brief Title: High-Dose Interferon Alfa and Interleukin-2 in Treating Patients With Metastatic Kidney Cancer or Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Collaborators: Cancer Biotherapy Research Group (Other)
Responsible Party: Robert O. Dillman, MD, Hoag Memorial Hospital Presbyterian
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065795; CBRG-9509; NBSG-9509; NCI-V97-1346
Record Dates: First submitted 1999-11-01; First posted 2004-07-07 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Kidney Cancer; Melanoma (Skin)
Keywords: stage IV renal cell cancer; recurrent renal cell cancer; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Carcinoma, Renal Cell | interventions — aldesleukin; Interferon-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon alfa

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells. Interleukin-2 may stimulate a person's white blood cells to kill kidney cancer or melanoma cells.

PURPOSE: Phase II trial to study the effectiveness of high-dose interferon alfa and interleukin-2 in treating patients with metastatic kidney cancer or melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety, efficacy, and antitumor activity of high dose interferon alfa-2b and interleukin-2 in patients with metastatic renal cell carcinoma or melanoma. II. Determine the toxic effects of interferon alfa-2b and interleukin-2 in these patients.

OUTLINE: This is an open label study. Patients receive subcutaneous interferon alfa-2b on days 1-4. Patients are hospitalized and receive bolus infusions of interleukin-2 (IL-2) followed by a continuous infusion on days 5-7. Patients are observed at least 12 hours following IL-2 treatment. Treatment is repeated every 4 weeks until disease progression or up to a maximum of six cycles. Patients are followed every 2 months for one year, then for survival.

PROJECTED ACCRUAL: If at least 1 response is seen in the first 14 patients in each group, a maximum of 40 patients per group will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven metastatic renal cell carcinoma or melanoma Measurable or evaluable disease No active brain metastases Previously treated CNS metastases responding to therapy are eligible, but CNS cannot be the site of evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: ECOG 0-2 Life Expectancy: Not specified Hematopoietic: Hematocrit at least 25 WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 PT and PTT within normal limits Hepatic: Bilirubin less than 2.0 mg/dL Renal: Creatinine less than 2.0 mg/dL Cardiovascular: No myocardial infarction within 6 months No medication for congestive heart failure or cardiac arrhythmias No hypertension (unless blood pressure is stable off medication) Pulmonary: Must have reasonable respiratory reserves and not require supplemental oxygen No dyspnea at rest Oxygen saturation must be greater than 90% for patients with risk of respiratory symptoms Other: Not HIV positive Not positive for hepatitis B antigen No chronic underlying immunodeficiency No concurrent active infection requiring antibiotic therapy Not pregnant or nursing No concurrent serious illness No family history of malignant hyperthermia No hypersensitivity to interferon alfa-2b and interleukin-2

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior interleukin-2 and interferon alfa-2b in combination therapy Chemotherapy: No prior systemic chemotherapy within 4 weeks of study and recovered Endocrine therapy: No concurrent corticosteroid therapy Radiotherapy: No prior radiotherapy within 4 weeks of interleukin-2 therapy No prior stereotactic radiosurgery or gamma knife therapy within 1 week of interleukin-2 therapy Surgery: No prior organ allograft transplantation Must be recovered from prior surgery Other: No concurrent cyclosporin therapy No concurrent treatment with other anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1996-01; Primary Completion 2000-01 (Actual); Study Completion 2000-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Dillman, MD, FACP, Study Chair — Cancer Biotherapy Research Group
Locations (4):
- United States (4):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Bloomington Hospital, Bloomington, Indiana
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - St. Joseph Regional Cancer Center, Bryan, Texas

REFERENCES:
- [Result] Dillman RO, Wiemann MC, Tai DF, Depriest CB, Soori G, Stark JJ, Mahdavi K, Church CK. Phase II trial of subcutaneous interferon followed by intravenous hybrid bolus/continuous infusion interleukin-2 in the treatment of renal cell carcinoma: final results of Cancer Biotherapy Research Group 95-09. Cancer Biother Radiopharm. 2006 Apr;21(2):130-7. doi: 10.1089/cbr.2006.21.130. PMID 16706633